CLINICAL TRIAL: NCT03102255
Title: The Effect of 'Sniffing Position & Nasal Tip Lifting' on the Pathway of Tracheal Tube in Nasal Cavity During Nasotracheal Intubation
Brief Title: The Effect of 'Sniffing Position & Nasal Tip Lifting' in Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical Professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20160707/26-2016-90/072
Record Dates: First submitted 2017-03-20; First posted 2017-04-05 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Intubation Complication
Keywords: Nasotracheal intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Performed nasotracheal intubation as usual. Sniffing position but doesn't lift a nasal tip.
  Interventions: Procedure: Sniffing position
- Nasal tip lifting (Experimental): Performed sniffing position and nasal tip lifting while the endotracheal tube insert patient's nasal cavity.
  Interventions: Procedure: Sniffing position; Procedure: Nasal tip lifting

INTERVENTIONS:
Procedure: Sniffing position — All procedure is done under sniffing position.
Procedure: Nasal tip lifting — Before inserting the endotracheal tube to patient's nose, the researcher lift up the nose tip.
  Arms: Nasal tip lifting

SUMMARY:
The goal of this prospective randomized study is to compare the effect of nasal tip lifting during nasotracheal intubation.

The question the investigators are trying to answer is: If the nasal tip is tilted, will the E-tube be more likely to enter the lower passage during nasal intubation?

DETAILED DESCRIPTION:
There are three nasal turbinates inside the nasal cavities. Each nasal cavity is divided into four spaces from these nasal turbinates, but the two spaces separated by the upper nasal turbinate are too narrow to be clinically meaningful. So when performing nasotracheal intubation, the tube enters one of the two spaces in low part divided into the lower turbinate. The middle turbinate, unlike others, a large number of blood vessels and nerves are distributed. Therefore, less hemorrhage might occurs when the tracheal tube enters into the lower pathway below the lower turbinate because the tube would not scratching the middle turbinate.

The hypothesis of this study is that the method 'sniffing position and nasal tip lifting' increases possibility to enter into lower pathway when the tube enters the nasal cavity. The purpose of a present study was to investigate the effect of 'sniffing position & nose' on the intranasal route of the tube.

ELIGIBILITY:
Inclusion Criteria:

* The patients who need to nasotracheal intubation for surgery.

Exclusion Criteria:

* Who doesn't agree to enroll.
* Who has severe nasal deformities.
* Who has a problem to make sniffing position or nasal tip lifting
* Who has severe nasal bleeding history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with nasal endotraheal tube in the lowest nasal pathway. | Through study completion, an average of 1 year
  After the endotracheal intubation is completed, the experimenter confirms by a fiberoptic bronchoscope which path the endotracheal tube is located.

SECONDARY OUTCOMES:
Nasal bleeding | Through study completion, an average of 1 year
  After nasotracheal intubation, the researcher confirm there is nasal bleeding or not. And if bleeding observed, the experimenter would check the amount.
Intubation time | Through study completion, an average of 1 year
  Check the time from initiation of insertion of E-tube to finish passing nasal path and to finish intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Study Director — Seoul National University Boramae Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed-Nusrath A, Tong JL, Smith JE. Pathways through the nose for nasal intubation: a comparison of three endotracheal tubes. Br J Anaesth. 2008 Feb;100(2):269-74. doi: 10.1093/bja/aem350. Epub 2007 Dec 14. PMID 18083994
- [Background] Patiar S, Ho EC, Herdman RC. Partial middle turbinectomy by nasotracheal intubation. Ear Nose Throat J. 2006 Jun;85(6):380, 382-3. PMID 16866113
- [Background] Williams AR, Burt N, Warren T. Accidental middle turbinectomy: a complication of nasal intubation. Anesthesiology. 1999 Jun;90(6):1782-4. doi: 10.1097/00000542-199906000-00039. No abstract available. PMID 10360881
- [Background] Dost P, Armbruster W. Nasal turbinate dislocation caused by nasotracheal intubation. Acta Anaesthesiol Scand. 1997 Jun;41(6):795-6. doi: 10.1111/j.1399-6576.1997.tb04787.x. PMID 9241346
- [Background] Scamman FL, Babin RW. An unusual complication of nasotracheal intubation. Anesthesiology. 1983 Oct;59(4):352-3. doi: 10.1097/00000542-198310000-00016. No abstract available. PMID 6614546
- [Derived] Kim H, Lee JM, Lee J, Hwang JY, Chang JE, No HJ, Won D, Choi S, Min SW. Influence of Nasal Tip Lifting on the Incidence of the Tracheal Tube Pathway Passing Through the Nostril During Nasotracheal Intubation: A Randomized Controlled Trial. Anesth Analg. 2018 Dec;127(6):1421-1426. doi: 10.1213/ANE.0000000000003673. PMID 30044295